CLINICAL TRIAL: NCT05149807
Title: A Randomized, Double-Blind, Multi-Center Phase II/III Clinical Study of PD-L1 Antibody/TGF-βRII (SHR-1701) Plus Tegafur Gimeracil Oteracil Potassium and Oxaliplatin Versus Placebo Plus Tegafur Gimeracil Oteracil Potassium and Oxaliplatin as Perioperative Treatment in Subjects With Resectable Gastric Cancer or Gastroesophageal Junction Cancer
Brief Title: Clinical Study of SHR-1701 Plus Chemotherapy as Perioperative Treatment in Subjects With Gastric Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: R&d strategy adjustment
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1701-III-308
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-07

CONDITIONS: Perioperative Treatment in Subjects With Locally Advanced Resectable Gastric Cancer or Gastroesophageal Junction Cancer
MeSH Terms: interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: This is a multi-center phase II/III clinical study consisting of two stages: Stage I is a single-arm open-label phase II study to preliminarily explore the efficacy and safety of SHR-1701 plus S-1 and oxaliplatin; Stage II is a randomized, double-blind, multi-center phase III study of SHR-1701 plus S-1 and oxaliplatin versus placebo plus S-1 and oxaliplatin as perioperative treatment in subjects with resectable GC or GEJC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1701 + Tegafur Gimeracil Oteracil Potassium and Oxaliplatin (Experimental)
  Interventions: Drug: SHR-1701 injection
- Placebo + Tegafur Gimeracil Oteracil Potassium and Oxaliplatin (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1701 injection — SHR-1701 injection Tegafur Gimeracil Oteracil Potassium Oxaliplatin
  Arms: SHR-1701 + Tegafur Gimeracil Oteracil Potassium and Oxaliplatin
Drug: Placebo — Placebo Tegafur Gimeracil Oteracil Potassium Oxaliplatin
  Arms: Placebo + Tegafur Gimeracil Oteracil Potassium and Oxaliplatin

SUMMARY:
This is a multi-center phase II/III clinical study consisting of two stages: Stage I is a single-arm open-label phase II study to preliminarily explore the efficacy and safety of SHR-1701 plus S-1 and oxaliplatin mainly by the endpoint of pCR rate.

Stage II is a randomized, double-blind, multi-center phase III study of SHR-1701 plus S-1 and oxaliplatin versus placebo plus S-1 and oxaliplatin as perioperative treatment in subjects with resectable GC or GEJC. A total of 846 treatment naïve subjects will be enrolled, and primary endpoint of this stage is Independent Review Committee (IRC)-assessed EFS.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with GC or GEJC, histologically confirmed to be adenocarcinoma, and have no previous anti-tumor treatments for GC or GEJC.
2. Aged 18 or above, male or female.
3. Be suitable for (investigator's assessment) and planning to undergo neoadjuvant therapy + radical surgery with curative intent before entering into the study.
4. locally advanced Gastric Cancer or Gastroesophageal Junction Cancer confirmed by investigator.
5. Be able to provide tumor tissue blocks.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
7. Life expectancy of ≥ 6 months.
8. Have adequate organ and bone marrow functions.
9. Women without childbearing potential refer to post-menopausal women, or women who underwent bilateral oophorectomy with medical records. Male subjects and female subjects of childbearing potential must agree to take a medically approved contraceptive measure (refer to Appendix 4) during the study, within 3 months after the last dose of investigational product (SHR-1701), and within 9 months after the last dose of chemotherapy agents (S-1 and oxaliplatin); have a negative serum pregnancy test result within 3 days prior to the start of study treatment and not be breastfeeding.
10. Subjects must agree and have signed the informed consent form, be willing and able to follow the scheduled visits, study treatment, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Have known squamous cell carcinoma, undifferentiated carcinoma, or other histological types of gastric cancer, or adenocarcinoma mixed with gastric cancer of other histological types.
2. Have unresectable factors, including unresectable tumors or contraindications to surgery or refusal of surgery.
3. Have more than 20% weight loss within 2 months prior to enrollment or randomization.
4. Have previously received some treatments or medications including anti-tumor treatments.
5. Diagnosed with other malignant tumors within 5 years prior to enrollment.
6. Have any active, known, or suspected autoimmune disease.
7. Have clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment or randomization; have gastrointestinal perforation and/or gastrointestinal fistula within 6 months prior to enrollment or randomization; have arterial/venous thrombotic events within 6 months prior to enrollment or randomization.
8. Have major vascular disease within 6 months prior to enrollment or randomization.
9. Have severe, unhealed, or dehisced wounds and active ulcers or untreated fractures.
10. Have intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to enrollment or randomization.
11. Have interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic disease.
12. Have known allergies to the study drug or their excipients; have severe allergic reactions to other monoclonal antibodies.
13. Have HIV infection or known AIDS, active untreated hepatitis or co-infection with hepatitis B and C.
14. Have uncontrolled cardiac symptoms or disease:
15. Have received systemic antibiotics for ≥ 7 days within 4 weeks prior to enrollment or randomization, or have unexplained fever > 38.5 °C during screening or before the first dose.
16. Have known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
17. Have been screened for other clinical studies but failed the screening because PD-L1 expression did not meet the inclusion criteria or met the exclusion criteria; have participated in clinical studies of any other drugs, less than 4 weeks or 5 half-lives of the drug between the last dose of these study treatments and enrollment/randomization for this study (whichever is longer).
18. Have a known history of psychotropic substance abuse or drug abuse.
19. Have other severe physical or psychiatric disorders or laboratory abnormalities, which may increase the risk of participation in this study or interfere with the study results, or deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Phase II : Pathological Complete Response pCR rate. | Up to approximately 23 months
  pCR rate is defined as the proportion of subjects whose specimens (including primary lesion and lymph nodes) obtained during GC or GEJC radical surgery are pathologically assessed to be free of residual live tumor cells after neoadjuvant therapy.
Phase III : Event-free Survival (EFS) | Up to approximately 57 months
  EFS is defined as time from randomization to PD or death (whichever occurs first), detailed that tumor progression/recurrence or new lesion confirmed by RECIST v1.1 criteria or death due to any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS). | Up to approximately 57 months
  DFS is defined as time from R0 resection to PD or death (whichever occurs first), detailed that tumor recurrence or new lesion confirmed by RECIST v1.1 criteria or death due to any cause.
Preoperative Objective Response Rate (ORR). | Up to approximately 57 months
  Preoperative ORR is defined as proportion of enrolled or randomized subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) according to RECIST v1.1 criteria during neoadjuvant therapy period.
Major pathological response (MPR) rates. | Up to approximately 23 months
  MPR rate is defined as proportion of subjects whose primary lesion specimens obtained during GC or GEJC radical surgery are pathologically assessed to have < 10% residual live tumor cells relative to the primary tumor tissue (Becker grade 1a or 1b) after neoadjuvant therapy.
R0 resection rate | Up to approximately 23 months
  R0 resection rate is defined as proportion of subjects without gross or microscopic residual tumor (negative margin) after neoadjuvant therapy and GC or GEJC radical surgery.
Overall Survival (OS). | Up to approximately 57 months
  OS is defined as time from randomization to death of any cause.
Percentage of Participants Who Experience One or More Adverse Events (AEs). | Up to approximately 57 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who experience at least one AE will be presented.
30-day postoperative mortality. | Up to approximately 24 months
  30-day postoperative mortality is defined as proportion of subjects who died due to any reason within 30 days after radical surgery for GC.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Southern Medical University NanFang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Subei people's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Air Force Military University Tangdu Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided